CLINICAL TRIAL: NCT02535325
Title: A Phase I Study of Methoxyamine Combined With Chemo-Radiation for Locally Advanced Non-Squamous Non-Small Cell Lung Cancer
Brief Title: Methoxyamine Hydrochloride, Pemetrexed Disodium, Cisplatin, and Radiation Therapy in Treating Patients With Stage IIIA-IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-01408; NCI-2015-01408 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 5514; 9834 (Other: Case Western Reserve University); 9834 (Other: CTEP); P30CA043703 (NIH)
Record Dates: First submitted 2015-08-27; First posted 2015-08-28 (Estimated); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Locally Advanced Lung Non-Squamous Non-Small Cell Carcinoma; Stage III Lung Adenocarcinoma AJCC v7; Stage III Lung Large Cell Carcinoma AJCC v7; Stage III Lung Non-Small Cell Cancer AJCC v7; Stage IIIA Lung Adenocarcinoma AJCC v7; Stage IIIA Lung Large Cell Carcinoma AJCC v7; Stage IIIA Lung Non-Small Cell Cancer AJCC v7; Stage IIIB Lung Adenocarcinoma AJCC v7; Stage IIIB Lung Large Cell Carcinoma AJCC v7; Stage IIIB Lung Non-Small Cell Cancer AJCC v7; Stage IV Lung Adenocarcinoma AJCC v7; Stage IV Lung Large Cell Carcinoma AJCC v7; Stage IV Lung Non-Small Cell Cancer AJCC v7
MeSH Terms: conditions — Adenocarcinoma of Lung | interventions — Radiotherapy, Conformal; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Radiotherapy, Intensity-Modulated; methoxyamine; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pemetrexed, methoxyamine, cisplatin, RT) (Experimental): CYCLES 1-2: Patients receive pemetrexed disodium IV over 10 minutes and methoxyamine hydrochloride PO day 1; and cisplatin IV over 0.5-24 hours on day 3. Patients also undergo 3-D conformal RT or IMRT QD 5 days a week (3 days of week 1 and 4 days of week 4) for 30 fractions total.
  CYCLES 3-4: Beginning at least 10 days after RT completion, patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 0.5-24 hours on day 1.
  Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3-Dimensional Conformal Radiation Therapy; Drug: Cisplatin; Radiation: Intensity-Modulated Radiation Therapy; Drug: Methoxyamine; Drug: Methoxyamine Hydrochloride; Drug: Pemetrexed; Drug: Pemetrexed Disodium

INTERVENTIONS:
Radiation: 3-Dimensional Conformal Radiation Therapy — Undergo 3-D conformal RT
  Other Names: 3-dimensional radiation therapy; 3D Conformal; 3D CONFORMAL RADIATION THERAPY; 3D CRT; 3D-CRT; Conformal Therapy; Radiation Conformal Therapy; Radiation, 3D Conformal
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Radiation: Intensity-Modulated Radiation Therapy — Undergo IMRT
  Other Names: IMRT; Intensity Modulated RT; Intensity-Modulated Radiotherapy; Radiation, Intensity-Modulated Radiotherapy
Drug: Methoxyamine — Given PO
  Other Names: TRC102 Base
Drug: Methoxyamine Hydrochloride — Given PO
  Other Names: TRC 102; TRC-102
Drug: Pemetrexed — Given IV
  Other Names: MTA; Multitargeted Antifolate; Pemfexy
Drug: Pemetrexed Disodium — Given IV
  Other Names: Alimta; Almita; LY231514; N-[4-[2-(2-Amino-4,7-dihydro-4-oxo-1H-pyrrolo[2,3-d]pyrimidin-5-yl)ethyl]benzoyl]-L-glutamic Acid Disodium Salt

SUMMARY:
This phase I trial studies the side effects and best dose of methoxyamine when given together with pemetrexed disodium, cisplatin, and radiation therapy in treating patients with stage IIIA-IV non-small cell lung cancer. Drugs used in chemotherapy, such as methoxyamine hydrochloride, pemetrexed disodium, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Radiation therapy uses high-energy x-rays to kill tumor cells and shrink tumors. Giving methoxyamine hydrochloride together with pemetrexed disodium, cisplatin, and radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of methoxyamine (TRC102) in combination with pemetrexed disodium (pemetrexed)-cisplatin and thoracic radiotherapy.

SECONDARY OBJECTIVES:

I. To (descriptively) assess the toxicity profile of methoxyamine (TRC102) in combination with pemetrexed-cisplatin and thoracic radiotherapy.

II. To (descriptively) assess the short-term progression-free survival at 6 months (PFS6) in the patients treated on this protocol.

III. To observe and record anti-tumor activity.

OUTLINE: This is a dose-escalation study of methoxyamine hydrochloride.

CYCLES 1-2: Patients receive pemetrexed disodium intravenously (IV) over 10 minutes and methoxyamine hydrochloride orally (PO) day 1; and cisplatin IV over 0.5-24 hours on day 3. Patients also undergo 3-dimensional (3-D) conformal radiation therapy (RT) or intensity-modulated radiation therapy (IMRT) once daily (QD) 5 days a week (3 days of week 1 and 4 days of week 4) for 30 fractions total.

CYCLES 3-4: Beginning at least 10 days after RT completion, patients receive pemetrexed disodium IV over 10 minutes and cisplatin IV over 0.5-24 hours on day 1.

Treatment repeats every 21 days for 4 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 weeks and then every 3 months for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologic diagnosis of adenocarcinoma or large cell carcinoma of the lung with confirmation by immunohistochemistry (e.g., transcription termination factor 1 [TTF-1] positivity) (histologic tissue diagnosis is recommended, but cytology is acceptable); stage IIIA/IIIB or oligometastatic stage IV in which the patient is still considered an appropriate candidate for aggressive chemoradiotherapy for the primary tumor; oligometastatic disease is defined as =< 5 metastatic sites (=< 3 lesions per organ); for intracranial metastasis, the patient should have asymptomatic disease that is stable on steroids or 1 to 3 symptomatic metastatic lesions treated with stereotactic radiosurgery (SRS)
* Eastern Cooperative Oncology Group (ECOG) performance status < 2
* Life expectancy of greater than 12 months
* Ability to swallow and retain orally-administered medication and does not have any clinically significant gastro-intestinal abnormalities (e.g., malabsorption syndrome or major resection of the stomach or bowel)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits OR
* Creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Hemoglobin >= 9 g/dL without transfusion within 7 days prior to enrollment
* The effects of methoxyamine (TRC102) on the developing human fetus are unknown; for this reason and because methoxyamine as well as other therapeutic agents used in this trial are known to be teratogenic. women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men and women treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of methoxyamine administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had prior chemotherapy or any other investigational drug within 30 days of registration or prior radiotherapy to the study treatment volume; prior surgery is allowed; there must be at least 6 weeks between mitomycin or nitrosoureas and any new therapy
* Patients who are receiving any other investigational agents
* Patients with a history of any active malignancy requiring on-going treatment, except basal cell carcinoma or squamous cell carcinoma of the skin
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to methoxyamine or to pemetrexed or cisplatin
* Undetectable haptoglobin or evidence of glucose-6-phophate dehydrogenase (G6PD) deficiency, pyruvate kinase deficiency, hemoglobinopathy, hereditary spherocytosis, thalassemia or other disorder associated with hemolysis
* Patients receiving any medications or substances that are inhibitors or inducers of nonsteroidal anti-inflammatory drugs (NSAIDS), probenecid, salicylates, sulfonamides are ineligible; concomitant drugs that are sensitive CYP450 substrates or strong and moderate CYP450 inducers and inhibitors should be avoided; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because methoxyamine is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with methoxyamine, breastfeeding should be discontinued if the mother is treated with methoxyamine; these potential risks may also apply to other agents used in this study
* Patients who are known to be human immunodeficiency positive (HIV)-positive and are on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with methoxyamine, pemetrexed or cisplatin; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of methoxyamine in combination with pemetrexed disodium, cisplatin, and radiation therapy | 21 days
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. MTD is defined as the highest dose level in which 0/6 or 1/6 patients suffer dose-limiting toxicity.
Incidence of toxicity of the combination therapy | Up to 6 months
  Will be graded according to NCI CTCAE version 5.0. Toxicity data will be tabulated.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | At 6 months
  PFS is analyzed using the Kaplan-Meier method. Factors, such as age, gender, baseline histology and lab correlates including uracil deoxyribonucleic acid (DNA) N-glycosylase (UNG), thymidylate synthase (TS), excision repair cross-complementation group 1 (ERCC1), Ki-67 and Topoisomerase II-alpha (TopoII-alpha) that predict survival will be identified by Cox model or extended Cox model.
Disease-free survival | Up to 6 months
  Disease-free survival is analyzed using the Kaplan-Meier method. Factors, such as age, gender, baseline histology and lab correlates including UNG, TS, ERCC1, Ki-67 and TopoII-alpha that predict survival will be identified by Cox model or extended Cox model.
Response rate (clinical/tumor response) | Up to 6 months
  The true response rate of the combination therapy for this patient population will be estimated based on the number of responses using a binomial distribution and its confidence intervals will be estimated using Wilson's method. The factors that predict the response will be identified by logistic regression.
Change in lab correlative expression levels (including UNG, TS, ERCC1, Ki-67 and TopoII-alpha) | Baseline to up to 6 months
  The change of lab correlatives measured at baseline and post-treatment will be compared by paired T-test for interval scale measure and McNemar test for nominal measure.

CONTACTS AND LOCATIONS:
Overall Officials: Tithi Biswas, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States